CLINICAL TRIAL: NCT01570595
Title: A Pilot Study of Positively Smoke Free on the Web (PSFW) for HIV-infected Smokers
Brief Title: Positively Smoke Free on the Web (PSFW) for Smokers Living With HIV
Acronym: PSFW
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: Albert Einstein College of Medicine (Other); University of Michigan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3358936; R21CA163100 (NIH)
Record Dates: First submitted 2012-03-14; First posted 2012-04-04 (Estimated); Last update posted 2014-05-12 (Estimated); Status verified 2014-05

CONDITIONS: Tobacco Use Cessation; Tobacco Cessation; Tobacco Use Disorder; Tobacco Dependence; Tobacco-Use Disorder; Virus, Human Immunodeficiency
Keywords: Tobacco Use Cessation; Tobacco Cessation; Tobacco Use Disorder; Tobacco Dependence; Tobacco-Use Disorder; Virus, Human Immunodeficiency
MeSH Terms: conditions — Tobacco Use Cessation; Tobacco Use Disorder; Acquired Immunodeficiency Syndrome | interventions — Standard of Care

ARMS (2):
- Web-Based Intervention (Experimental): This group will be asked to participate in the online quit smoking program. At their first visit, they will be given an ID number to log in to the quit smoking program, and they will complete their first log in with the research assistant. The online program is made up of 8 separate online sessions that are supposed to be completed approximately once per week. Each sessions is written to take an average reader 15-30 minutes to complete. The entire program is meant to be completed in 7 weeks. At the first visit, participants are asked to provide an email address and/or cell phone number so reminders can be sent, by email or text message, to complete the sessions. If participants are late completing a session, they may receive call from clinic staff as a reminder.
  Interventions: Behavioral: Web-Based Tailored Smoking Cessation Intervention
- Standard Care (Active Comparator): This group will receive "standard care" for their smoking, including advice to quit, a quit-smoking brochure, and an offer of three months of nicotine replacement therapy (nicotine patches).
  Interventions: Behavioral: Web-Based Tailored Smoking Cessation Intervention; Behavioral: Standard of Care

INTERVENTIONS:
Behavioral: Web-Based Tailored Smoking Cessation Intervention — The Experimental group will be given an ID number to log in to the quit smoking program, and complete their first log-in with a research assistant. The online program is made up of 8 separate, weekly online sessions that take approximately 15-30 minutes to complete. The entire program is meant to be completed in 7 weeks. Participants are asked to provide an email address and/or cell phone number so reminders can be sent to complete the sessions. If participants are late completing a session, they will receive a call from clinic staff as a reminder. The "standard care" group will receive advice to quit, a quit-smoking brochure, and an offer of three months of nicotine replacement therapy (nicotine patches).
  Other Names: Tailored Cessation; Web-Based Intervention; Web-Based Cessation
Behavioral: Standard of Care — advice to quit, a quit-smoking brochure, and an offer of three months of nicotine replacement therapy (nicotine patches).
  Arms: Standard Care

SUMMARY:
The purpose of this study is to evaluate the first web-based cessation program developed expressly for people living with HIV who smoke tobacco. Main study goals are (1) to evaluate the website's feasibility (i.e., recruitment, adherence, retention, and satisfaction) and (2) to complete a prospective, randomized controlled trial comparing the efficacy of the online program to standard care with a primary outcome of 3 month point-prevalence abstinence.

DETAILED DESCRIPTION:
Positively Smoke Free on the Web is the first web-based cessation program developed expressly for people living with HIV (PLWH) who smoke tobacco. It is a resource that is ready for clinical use, but its feasibility and efficacy have yet to be studied. Main study goals are (1) to evaluate the website's feasibility (i.e., recruitment, adherence, retention, and satisfaction) in a cohort of 69 PLWH smokers, and (2) to complete a prospective, randomized controlled trial comparing the efficacy of the online program to standard care (total N = 138) with a primary outcome of 3 month point-prevalence abstinence.

ELIGIBILITY:
Inclusion Criteria:

* Laboratory confirmation of HIV infection
* Montefiore Medical Center Infectious Disease Clinic patient
* Current tobacco user
* Affirmed motivation to quit within the next 6 months
* Have home access to the Internet
* Read above 4th grade level (by REALM)
* Willingness to grant informed consent and undergo randomization

Exclusion Criteria:

* Pregnant or breastfeeding women
* People with contraindications to nicotine replacement therapy
* People currently receiving other tobacco treatment
* Spouses, partners, and/or roommates of current study participants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2011-09; Primary Completion 2013-07 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
24-hour Point-prevalence tobacco abstinence | 3 months
  The proportion of each group achieving 24-hour point prevalence abstinence at Visit 3 (i.e., abstinence on or around Day 121 - 3 months post-Quit Day in the Intervention condition) by exhaled carbon monoxide, an accepted method for biochemical validation of abstinence.

SECONDARY OUTCOMES:
Degree of Participation in Intervention (Feasibility) | 3 Months (duration of intervention)
  Intervention feasibility will be assessed using variables such as total # of logins, # of sessions viewed, # of web pages viewed, # of mouse clicks on interactive features, total time logged on to the site (automatic logoff occurs after 30 minutes of inactivity), proportion completing the final study visit, program satisfaction survey results, and total # of reminder phone calls/texts placed by clinic staff.
Knowledge and Behavior Change | Day 0, 42, 121
  Validated measures will be used to collect data on continuous abstinence, number of quit attempts, and current daily cigarette consumption. Composite quit indices will be analyzed, especially the combination of 3 month continuous abstinence with expired carbon monoxide (ECO) confirmation. We will also analyze results of validated measures that have known associations with cessation outcomes (tobacco knowledge, depression, anxiety, motivation to quit, self-concept, perceived risks/benefits, self-efficacy, and decisional balance).

CONTACTS AND LOCATIONS:
Locations (1):
- Albert Einstein College of Medicine of Yeshiva University, The Bronx, New York, United States

REFERENCES:
- [Derived] Shuter J, Pearlman BK, Stanton CA, Moadel AB, Kim RS, Weinberger AH. Gender Differences among Smokers Living with HIV. J Int Assoc Provid AIDS Care. 2016 Sep;15(5):412-7. doi: 10.1177/2325957416649439. Epub 2016 May 23. PMID 27215559
- [Derived] Shuter J, Morales DA, Considine-Dunn SE, An LC, Stanton CA. Feasibility and preliminary efficacy of a web-based smoking cessation intervention for HIV-infected smokers: a randomized controlled trial. J Acquir Immune Defic Syndr. 2014 Sep 1;67(1):59-66. doi: 10.1097/QAI.0000000000000226. PMID 25118794
- See also: Positively Smoke Free Website — http://www.positivelysmokefree.org